CLINICAL TRIAL: NCT05044000
Title: Effect of Deep Propioceptive Stimulation on Sleep Disorders, Behavior and Brain Connectivity in Adults with Prader-Willi Syndrome
Brief Title: Effect of Deep Propioceptive Stimulation in Prader-Willi Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Assumpta Caixas, Principal investigator, Corporacion Parc Tauli
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Endocrinology Parc Tauli; PI21/00459 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2021-08-31; First posted 2021-09-14 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Sleep Disorder; Hyperphagia; Behavior Disorders
MeSH Terms: conditions — Sleep Wake Disorders; Hyperphagia; Mental Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Heavy blanket and similar blanket (not heavy)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heavy blanket (Experimental): Patients will start with heavy blanket during 15 days
  Interventions: Device: Deep propioceptive stimulation
- Non-heavy blanket (Placebo Comparator): Patients will start with non-heavy blanket during 15 days
  Interventions: Device: Deep propioceptive stimulation

INTERVENTIONS:
Device: Deep propioceptive stimulation — Participants will start using the blanket (of the arm name), 30 days wash-out and 15d with the other blanket

SUMMARY:
The main objective is to study the effect of deep propioceptive stimulation with a heavy blanket for 2 weeks compared with a placebo blanket on sleep quality and behavior in patients with PWS

DETAILED DESCRIPTION:
Prader-Willi syndrome (PWS) is a genetic disease associated with sleep disorders whose etiology is partly central due to the inherent hypothalamic deficit. It is associated with low cognitive performance and worsening behavior with more impulsivity, tantrums, scratches and obsession for food. Deep propioceptive stimulation with a heavy blanket (HB) stimulates the parasympathetic system and improves the state of anxiety in persons with autism or other causes of intellectual disability and/or psychopathology. To date, there are no studies evaluating the effect of HB on sleep quality or brain activity in persons with PWS. The main objective is to study the effect of HB for 2 weeks compared to a placebo blanket on sleep quality and behavior in patients with SPW.

Methodology: Actigraphy, questionnaires, crossover study in 60 patients with PWS, with HB/placebo blankets (15 days each). Effect of HB on brain connectivity with functional magnetic resonance imaging in 30 patients and 30 controls. Expected results: PWS group will show worse sleep quality and behavior that will improve after using HB. Brain connectivity will be different with/without HB. These favorable changes will help to justify the use of this ecological treatment and its inclusion in the NHS clinical practice guidelines for improving the quality of life of these patients and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PWS genetically confirmed at least 16y old willing to participate and being able to be still in the MRI.

Exclusion Criteria:

1. Age < 16 years old
2. Presence of uncontrolled Obstructive Sleep Apnea (Residual AHI ≥ 30).
3. Narcolepsy or other sleep disorders with daily somnolence
4. Intolerance to the heavy blanket in spite of previous adaptation sessions
5. Active psychopathological disorder that may interfere with sleep
6. Use of hypnotic or sleep regulator drugs (change of dose in the last 3 months)
7. Contraindications for MRI
8. Impossibility to stay still during MRI adquisition

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Changes in number of awakenings | 14 nights
  measured by actigraphy
Change in duration of awakenings | 14 nights
  minutes measured by actigraphy

SECONDARY OUTCOMES:
Number of tantrums | 15 days
  caregivers report
number of skin injuries | 15 days
  physical examination by the principal investigator or collaborators
Interest for food | 15 days
  Hyperphagia questionnaire for clinical trials (9 items from 1-4, maximum score 36, more is worse)
Brain connectivity | 1 day
  functional magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Assumpta Caixas, MD, PhD, Principal Investigator — Corporacio Sanitaria Parc Tauli
Locations (1):
- Consorci Corporacio Sanitaria Parc TAuli, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No